CLINICAL TRIAL: NCT01785082
Title: Prospective, Randomized, Controlled, Multi-centric, Phase III Study for the Early Identification of Low-risk Patients After Partial Liver Resection by the LiMAx-test
Brief Title: Fast-track LiveR: Study for the Early Identification of Low-risk Patients After Partial Liver Resection by the LiMAx-test
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Humedics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM-001
Record Dates: First submitted 2013-01-25; First posted 2013-02-07 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Liver Failure
Keywords: 13-C-Methacetin; partial liver resection; liver function tests
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LiMAx-group (Experimental): Intravenous pre- and post-surgical injection of 0.4% 13-C-Methacetin solution. Dosage is adapted due to body weight (2 mg/kg). A LiMAx-test of >150 µg/kg/h would correspond to a general ward indication.
  Interventions: Drug: 13-C-Methacetin
- control group (No Intervention): Control group without intervention. Post-surgical management as defined prior to surgery following well-established clinical standards.

INTERVENTIONS:
Drug: 13-C-Methacetin — intravenous injection of 0.4% 13-C-Methacetin solution, once before partial liver resection, once after partial liver resection
  Arms: LiMAx-group

SUMMARY:
The purpose of this study is to investigate safety and efficacy of intravenously injected 0.4% 13-C-Methacetin solution for the determination of liver function with the LiMAx-test on patients with partial liver resection. The LiMAx-test is compared with an untreated control group and post-surgical management of both groups is investigated.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients of 18 years or older which are able to give informed consent with indication for surgical partial liver resection according to OPS code 5-502; this includes benign and malign tumors.
* patients with pre-surgical thin-layer CT or MRT of the liver not older than 6 weeks or patients where a pre-surgical thin-layer CT or MRT of the liver is planned before surgery.
* written informed consent

Exclusion Criteria:

at screening:

* anamnestic known hypersensitivity against one of the study drugs, their ingredients or drugs with chemically similar structure (in particular paracetamol)
* participation in another clinical trials within 4 weeks before inclusion
* patients with previous liver surgery (OPS-Code 5-502), including biliodigestive anastomosis, excluding cholecystectomy.
* patients which underwent interventions such as radiofrequency ablation, biopsies or smaller surgeries within 6 weeks before inclusion
* patients anticipated for biliodigestive anastomosis and/or suffering from a Klatskin-tumor
* patients with a ASA (American Society of Anesthesiologists) classification >3
* patients anticipated for laparoscopic partial liver resection
* patients which are intended to be simultaneously treated with an interventional technique (e.g. radio frequency ablation RFA, embolization)
* patients which are intended to simultaneously get a surgery on other organs (excluding cholecystectomy)
* patients which are intended to simultaneously get a vascular anastomosis (e.g. portal vein resection)
* patients with known hepatic cirrhosis or known severe fibrosis (e.g. Ishak-score grade >4)
* patients with congenital metabolic diseases, in particular hepatic storage diseases
* hepatic infection with Echinococcus multilocularis
* patients with known non-infectious, auto-immune conditioned chronic inflammatory diseases (e.g. autoimmune hepatitis, Morbus Crohn, colitis ulcerativa)
* patients with severe cardiovascular diseases and/or severe diseases of the respiratory system which receive intensive care in any case (e.g. heart surgery, bypass surgery, cardiac valve replacement, unstable angina pectoris, severe coronary heart disease with intervention during the last 6 months, severe COPD (chronic obstructive pulmonary disease), severe asthma with concomitant cortisone medication)
* patients with severe bacterial infection at screening
* patients with known immunodeficiency
* heavy smokers (>20 cigarettes a day)
* patients which are unable to understand the study and its possible implications because of addiction or other diseases
* patients who are suspected not to cooperate or to comply to the trial protocol
* patients accommodated in an institution due to public or legal authority
* pregnant or lactating women
* women with child-bearing potential, excluding: negative pregnancy test and commitment to be sexually inactive until day 30 after surgery or discharge; postmenopause (12 months of natural occurring amenorrhoea); at least 6 weeks after ovariectomy with or without hysterectomy

at visit 2:

* patients anticipated for laparoscopic partial liver resection
* patients which are intended to be simultaneously treated with an interventional technique (e.g. radio frequency ablation RFA, embolization)
* patients which are intended to simultaneously get a surgery on other organs (excluding cholecystectomy)
* patients which are intended to simultaneously get a vascular anastomosis (e.g. portal vein resection)
* patients with known hepatic cirrhosis or known severe fibrosis (e.g. Ishak-score grade >4)
* hepatic infection with Echinococcus multilocularis
* patients with severe cardiovascular diseases and/or severe diseases of the respiratory system which receive intensive care in any case (e.g. heart surgery, bypass surgery, cardiac valve replacement, unstable angina pectoris, severe coronary heart disease with intervention during the last 6 months, severe COPD (chronic obstructive pulmonary disease), severe asthma with concomitant cortisone medication)
* patients anticipated for biliodigestive anastomosis and/or suffering from a Klatskin-tumor
* patients with a ASA (American Society of Anesthesiologists) classification >3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
number of correctly determined positive patients in each trial group | no later than day 30 after surgery
  Correctly determined positive patients are patients which are transferred to general ward after surgery because of the result of the LiMAx-test (LiMAx-group) or general diagnosis (control group). Patients have to stay at general ward until discharge no later than day 30 after surgery.

SECONDARY OUTCOMES:
number of incorrectly determined positive patients in each trial group | no later than day 30 after surgery
  Incorrectly determined positive patients are patients which are transferred to general ward after surgery because of the result of the LiMAx-test or general diagnosis (control group) and do not stay at general ward until discharge or are discharged later than 30 days after surgery.
sensitivity | 1 year after trial start (anticipated December 2013)
  number of correctly predicted positive patients / (number of correctly predicted positive patients + number of incorrectly predicted negative patients)
specificity | 1 year after trial start (anticipated December 2013)
  number of correctly predicted negative patients / (number of correctly predicted negative patients + number of incorrectly predicted positive patients)
positive predictive value (PPV) | 1 year after trial start (anticipated December 2013)
  number of correctly predicted positive patients / (number of correctly predicted positive patients + number of incorrectly predicted positive patients)
negative predictive value (NPV) | 1 year after trial start (anticipated December 2013)
  number of correctly predicted negative patients / (number of correctly predicted negative patients + number of incorrectly predicted negative patients)
mortality | 1 year after trial start (anticipated December 2013)
  total mortality until day 30 post-surgical
number of patients with post-surgical liver failure (PHLF) | 1 year after trial start (anticipated December 2013)
  PHLF according to the Rahbari-Score
total number of complications | 1 year after trial start (anticipated December 2013)
  total number of complications of grade IIIa (surgical, endoscopic or radiological intervention) to grade V (death)
changes of routine laboratory data | until day 30 after surgery
  assessment of clinical data (sodium, potassium, creatinine, urea, protein, albumin, total bilirubin, AST, ALT, AP, GGT, blood count, INR, PTT). In addition, clinical data as pulse or blood pressure are recorded.

OTHER OUTCOMES:
pre- and post-surgical volumetric analysis of the liver | immediately pre and post surgery
  Pre-surgical volumetric analysis of liver and tumor by CT or MRT and post-surgical volumetric analysis of the resected liver.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Stockmann, PD Dr. med., Principal Investigator — Dept. of General-, Visceral- and Graft Surgery, Charité Campus Virchow-Hospital, Augustenburger Platz 1, 13353 Berlin, Germany
Locations (4):
- Germany (4):
  - Dept. of General-, Visceral- and Graft Surgery, Charité Campus Virchow-Hospital, Berlin
  - Dept. of General- and Visceral Surgery, Jena University Hospital, Jena
  - Clinic and Policlinic for Visceral-, Graft-, Thorax- and Vascular Surgery, Leipzig University Hospital, Leipzig
  - Clinic and Policlinic for General- Visceral- and Graft Surgery, Würzburg University Hospital, Würzburg

REFERENCES:
- [Result] Stockmann M, Vondran FWR, Fahrner R, Tautenhahn HM, Mittler J, Bektas H, Malinowski M, Jara M, Klein I, Lock JF; Collaborative Fast-track Liver Study Group. Randomized clinical trial comparing liver resection with and without perioperative assessment of liver function. BJS Open. 2018 Jun 14;2(5):301-309. doi: 10.1002/bjs5.81. eCollection 2018 Sep. PMID 30263981
- See also: EU clinical trials register with results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2010-023095-31/results